CLINICAL TRIAL: NCT02060006
Title: A Double-Blind Randomized Placebo Controlled Trial for Prevention of Tuberculosis-Immune Reconstitution Inflammatory Syndrome With Non-Steroid Anti-Inflammatory Drugs (NSAIDs) in HIV-Infected Adults
Brief Title: TB-IRIS NSAID Cox-2 Inhibitor Prevention Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Stellenbosch (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Prof Jean Nachega, Professor Extraordinary, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO13060453
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Tuberculosis
Keywords: TB; IRIS
MeSH Terms: conditions — Tuberculosis | interventions — Meloxicam; Cyclooxygenase 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo 7.5 mg daily for 8 weeks (Placebo Comparator): Placebo 7.5 mg once-daily First 8 weeks of ART Only Control arm
- Meloxicam 7.5 mg once-daily (Experimental): Meloxicam 7.5mg once-daily for 8 weeks
  Interventions: Drug: Meloxicam 7.5mg daily for 8 weeks

INTERVENTIONS:
Drug: Meloxicam 7.5mg daily for 8 weeks — Meloxicam 7.5mg daily for 8 weeks
  Other Names: Cox-2 Inhibitor
  Arms: Meloxicam 7.5 mg once-daily

SUMMARY:
Background: Non-Steroid Anti-Inflammatory Drugs (NSAIDs) reduce pain and inflammation by inhibiting cyclooxygenase, an enzyme in the pathway for formation of prostaglandins and thromboxane. Prior studies have proven the role of ibuprofen (an NSAID) in modulating lung injury and decreasing pulmonary damage in cystic fibrosis. While there has been an intense effort by the scientific community to define the best treatment strategies for tuberculosis immune reconstitution inflammatory syndrome (TB-IRIS), to our knowledge there is no available study evaluating preventive strategies using anti-inflammatory agents for TB-IRIS, a highly morbid complication in HIV-infected TB patients initiating antiretroviral therapy (ART).

Design and Methods: We propose to conduct a single center double-blind placebo-controlled randomized trial to investigate the efficacy of daily self-administered Meloxicam (a NSAID) versus placebo for prevention of Tuberculosis associated Immune Reconstitution Inflammatory Syndrome (TB-IRIS). A total of 150 HIV-infected adults who are treated for Tuberculosis for at least 2 weeks and about to initiate HIV treatment at Brewelskloof Hospital, Worcester, and Tygerberg Teaching Hospital, Cape Town, will be randomized to one of the following treatments: Meloxicam 7.5 mg tablet once-a-day, the experimental arm, versus Placebo tablet once-a-day, the control arm, for 8 weeks. All patients will be followed up for 12 months. Primary efficacy outcome: The decrease of the incidence of paradoxical TB IRIS by at least 20%; Primary safety outcome: The proportion of patients who temporarily or permanently discontinue Meloxicam due to any adverse event (e.g. dyspepsia or gastro-intestinal upset). Secondary outcomes are: 1) the proportion of patients in each arm with the following indicators of TB-IRIS severity/quality of life (QOL) (degree of pain or discomfort >III, presence of local or disseminated suppuration/abscess of any site, unscheduled clinic visits, hospitalizations, missed more than a day at work, etc; 2) The incidence of other types of IRIS (e.g. Kaposi Sarcoma or cryptococcal meningitis).

This study will provide important and novel data on the feasibility and efficacy of using a cheap, widely available NSAID used in both developed and developing countries, as a preventive intervention for TB-IRIS that could be quickly put into practice if proven to be effective

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females age 18 years of age or older
* Evidence of HIV-1 infection
* TB treatment (<2 weeks) and initiating EFV-based antiretroviral therapy as per the South African Department of Health Guidelines
* Living in the study site catchment area and having had a known address for more than 3 months
* Written informed consent

Exclusion Criteria:

* History of aspirin sensitivity and allergies to other NSAIDs
* Current or recent use (<3 months) of aspirin, NSAIDs, or anticoagulants such as warfarin.
* Current or recent use of corticosteroid therapy
* History of gastro-intestinal bleeding or peptic ulcer
* History of cardiovascular thrombotic events (myocardial infarction or stroke), hypertension, or congestive heart failure
* Severe renal impairment as evidenced by creatinine clearance <50 (Cockcroft- Gault Formula)
* Severe liver disease (ALT > five times upper limit of normal)
* Presence of a medical condition likely to result in death within 6 months from start of ART. These conditions include suspected or CNS lymphoma, PMLE and disseminated visceral Kaposi's sarcoma
* Cognitive disorder(s) that could impair ability to comply with study requirements, as determined by the study physician
* Karnofsky performance score <60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04

PRIMARY OUTCOMES:
Incidence of TB IRIS | 6 months

SECONDARY OUTCOMES:
Proportion discontinuing Meloxicam due to adverse event | 6 months
The proportion of patients in each arm with the following indicators of TB-IRIS severity/quality of life (QOL) (degree of pain or discomfort >III | 6 months
The proportion of patients with local or disseminated suppuration/abscess of any site, unscheduled clinic visits, hospitalizations, missed more than a day at work, etc | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stellenbosch University Tygerberg Hospital, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Eshun-Wilson I, Havers F, Nachega JB, Prozesky HW, Taljaard JJ, Zeier MD, Cotton M, Simon G, Soentjens P. Evaluation of paradoxical TB-associated IRIS with the use of standardized case definitions for resource-limited settings. J Int Assoc Physicians AIDS Care (Chic). 2010 Mar-Apr;9(2):104-8. doi: 10.1177/1545109710361537. Epub 2010 Feb 16. PMID 20160249
- [Background] Meintjes G, Wilkinson RJ, Morroni C, Pepper DJ, Rebe K, Rangaka MX, Oni T, Maartens G. Randomized placebo-controlled trial of prednisone for paradoxical tuberculosis-associated immune reconstitution inflammatory syndrome. AIDS. 2010 Sep 24;24(15):2381-90. doi: 10.1097/QAD.0b013e32833dfc68. PMID 20808204
- [Background] Meintjes G, Lawn SD, Scano F, Maartens G, French MA, Worodria W, Elliott JH, Murdoch D, Wilkinson RJ, Seyler C, John L, van der Loeff MS, Reiss P, Lynen L, Janoff EN, Gilks C, Colebunders R; International Network for the Study of HIV-associated IRIS. Tuberculosis-associated immune reconstitution inflammatory syndrome: case definitions for use in resource-limited settings. Lancet Infect Dis. 2008 Aug;8(8):516-23. doi: 10.1016/S1473-3099(08)70184-1. PMID 18652998
- [Background] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray A, Gengiah T, Nair G, Bamber S, Singh A, Khan M, Pienaar J, El-Sadr W, Friedland G, Abdool Karim Q. Timing of initiation of antiretroviral drugs during tuberculosis therapy. N Engl J Med. 2010 Feb 25;362(8):697-706. doi: 10.1056/NEJMoa0905848. PMID 20181971
- [Background] Blanc FX, Sok T, Laureillard D, Borand L, Rekacewicz C, Nerrienet E, Madec Y, Marcy O, Chan S, Prak N, Kim C, Lak KK, Hak C, Dim B, Sin CI, Sun S, Guillard B, Sar B, Vong S, Fernandez M, Fox L, Delfraissy JF, Goldfeld AE; CAMELIA (ANRS 1295-CIPRA KH001) Study Team. Earlier versus later start of antiretroviral therapy in HIV-infected adults with tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1471-81. doi: 10.1056/NEJMoa1013911. PMID 22010913
- [Background] Havlir DV, Kendall MA, Ive P, Kumwenda J, Swindells S, Qasba SS, Luetkemeyer AF, Hogg E, Rooney JF, Wu X, Hosseinipour MC, Lalloo U, Veloso VG, Some FF, Kumarasamy N, Padayatchi N, Santos BR, Reid S, Hakim J, Mohapi L, Mugyenyi P, Sanchez J, Lama JR, Pape JW, Sanchez A, Asmelash A, Moko E, Sawe F, Andersen J, Sanne I; AIDS Clinical Trials Group Study A5221. Timing of antiretroviral therapy for HIV-1 infection and tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1482-91. doi: 10.1056/NEJMoa1013607. PMID 22010914
- [Background] Konstan MW, Schluchter MD, Xue W, Davis PB. Clinical use of Ibuprofen is associated with slower FEV1 decline in children with cystic fibrosis. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1084-9. doi: 10.1164/rccm.200702-181OC. Epub 2007 Sep 13. PMID 17872492
- [Background] Kvale D, Ormaasen V, Kran AM, Johansson CC, Aukrust P, Aandahl EM, Froland SS, Tasken K. Immune modulatory effects of cyclooxygenase type 2 inhibitors in HIV patients on combination antiretroviral treatment. AIDS. 2006 Apr 4;20(6):813-20. doi: 10.1097/01.aids.0000218544.54586.f1. PMID 16549964